CLINICAL TRIAL: NCT02288312
Title: Food Effect and Dosage Form Proportionality Study of Eslicarbazepine Acetate Market Formulation in Healthy Volunteers
Brief Title: Food Effect and Dosage Form Proportionality Study of Eslicarbazepine Acetate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-117
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BIA 2-093 800 mg fasting (Experimental): Tablets 800 mg. Administration:Oral.
  Interventions: Drug: BIA 2-093
- BIA 2-093 800 mg fed (Experimental): Tablets 800 mg. Administration:Oral.
  Interventions: Drug: BIA 2-093
- BIA 2-093 400 mg (Experimental): Tablets 2 x 400 mg. Administration:Oral.
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate

SUMMARY:
Single-centre, open-label, randomised, gender-balanced, 3-way crossover, 3-period, 3-sequence study in 18 healthy male and female subjects.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, gender-balanced, 3-way crossover, 3-period, 3-sequence study in 18 healthy male and female subjects. The study consisted of 3 periods separated by a washout of 7 days or more between doses. Subjects received a single oral 800 mg dose of eslicarbazepine acetate following a standard meal in one period, and following at least 10 hours of fasting in two periods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 55 years, inclusive.
* Subjects of body mass index (BMI, kg/m2) within the normal range [4], i.e., between 18.50 and 24.99, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, and 12-lead ECG.
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission to first treatment period.
* Subjects who had negative tests for HBsAg, anti-HCVAb and anti- HIV-1 and HIV-2 Ab at screening.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening.
* Subjects who were non-smokers or ex-smokers who discontinued smoking at least 3 months prior to admission.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery (hysterectomy or tubal ligation) or, if of childbearing potential, she used one of the following methods of contraception: intrauterine device (by the study subject) + condom (by the partner), diaphragm (by the study subject) + condom (by the partner), or spermicide (by the study subject) + condom (by the partner).
* (If female) She had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, or
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who used medicines within 2 weeks of first admission that, in the opinion of the investigator, may affect the safety or other study assessments.
* Subjects who used any investigational drug or participated in any clinical trial within 2 months of their first admission.
* Subjects who had previously received eslicarbazepine acetate (ESL, BIA 2-093).
* Subjects who donated or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not used and approved effective contraceptive method or she used oral contraceptives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Period 1 - ESL 800 mg, in fasting (4 days) Period 2 - ESL 800 mg, in fed (4 days) Period 3 - ESL 800 mg (2x400mg), in fasting (4 days)
  Washout periods - 7 days between dosing days
- Group B: Period 1 - ESL 800 mg (2x400mg), in fasting (4 days) Period 2 - ESL 800 mg, in fasting (4 days) Period 3 - ESL 800 mg, in fed (4 days)
  Washout periods - 7 days between dosing days
- Group C: Period 1 - ESL 800 mg, in fed (4 days) Period 2 - ESL 800 mg (2x400mg), in fasting (4 days) Period 3 - ESL 800 mg, in fasting (4 days)
  Washout periods - 7 days between dosing days
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 6 | 6 | 6
Completed | 5 | 6 | 6
Not Completed | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence A: Period 1 - ESL 800 mg, in fasting Period 2 - ESL 800 mg, in fed Period 3 - ESL 800 mg (2x400mg), in fasting
- Sequence B: Period 1 - ESL 800 mg (2x400mg), in fasting Period 2 - ESL 800 mg, in fasting Period 3 - ESL 800 mg, in fed
- Sequence C: Period 1 - ESL 800 mg, in fed Period 2 - ESL 800 mg (2x400mg), in fasting Period 3 - ESL 800 mg, in fasting
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Sequence C | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cmax (BIA 2-005)
Description: Cmax (BIA 2-005) - maximum observed plasma drug concentration of BIA 2-005 (BIA 2-093 metabolite)
Time Frame: pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours postdose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 800 mg Fasting; BIA 2-093 800 mg Fed: Tablets 800 mg. Administration:Oral.
  BIA 2-093
- BIA 2-093 800 mg (2 x 400 mg): Tablets 2 x 400 mg. Administration:Oral.
  BIA 2-093
Arm/Group | BIA 2-093 800 mg Fasting | BIA 2-093 800 mg Fed | BIA 2-093 800 mg (2 x 400 mg)
Number analyzed (Participants) | 18 | 17 | 17
ng/mL | 10973 (2628) | 11044 (2495) | 11022 (2748)

2. Secondary Outcome: AUC0-t (BIA 2-005)
Description: AUC0-t (BIA 2-005) - the area under the plasma concentration-time curve from time zero to the last sampling time at which BIA 2-005 concentrations are at or above the limit of quantification, calculated by the linear trapezoidal rule (BIA 2-005 is a BIA 2-093 metabolite)
Time Frame: pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours postdose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 2-093 800 mg Fasting | BIA 2-093 800 mg Fed | BIA 2-093 800 mg (2 x 400 mg)
Number analyzed (Participants) | 18 | 17 | 17
ng.h/mL | 241651 (50381) | 234092 (50510) | 242375 (48599)

3. Secondary Outcome: Tmax (BIA 2-005)
Description: tmax (BIA 2-005) - the time of occurrence of Cmax of BIA 2-005 (BIA 2-005 is a BIA 2-093 metabolite)
Time Frame: pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours postdose.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIA 2-093 800 mg Fasting | BIA 2-093 800 mg Fed | BIA 2-093 800 mg (2 x 400 mg)
Number analyzed (Participants) | 18 | 17 | 17
hours | 2.64 (1.65) | 2.75 (2.31) | 2.56 (1.58)

4. Secondary Outcome: AUC0-∞ (BIA 2-005)
Description: AUC0-∞ (BIA 2-005) - the area under the plasma BIA 2-005 concentration versus time curve from time zero to infinity, calculated from AUC0-t + (Clast/λz), where Clast is the last quantifiable concentration and λz the apparent terminal rate constant; (BIA 2-005 is a BIA 2-093 metabolite)
Time Frame: pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours postdose.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 2-093 800 mg Fasting | BIA 2-093 800 mg Fed | BIA 2-093 800 mg (2 x 400 mg)
Number analyzed (Participants) | 18 | 17 | 17
ng.h/mL | 243808 (50464) | 236089 (50764) | 244821 (48873)

ADVERSE EVENTS:
Arm/Group | BIA 2-093 800 mg Fasting | BIA 2-093 800 mg Fed | BIA 2-093 800 mg (2 x 400 mg)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 3/18 | 2/17 | 2/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 800 mg Fasting (N=18) | BIA 2-093 800 mg Fed (N=17) | BIA 2-093 800 mg (2 x 400 mg) (N=17)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
CPK increased (Investigations) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other